CLINICAL TRIAL: NCT03351647
Title: Identification of Biological Predictive Factors of Clinical Response to Ustekinumab in Patients With Anti-Tumor Necrosis Factor (TNF) Antagonists Refractory Crohn's Disease: Interest of Dosage of C Reactive Protein (CRP), Calprotectin, Ustekinumab Through Levels and Antibodies
Brief Title: Predictive Factors of Clinical Response to Ustekinumab in Active Crohn's Disease
Acronym: SAFARI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0218
Record Dates: First submitted 2017-10-30; First posted 2017-11-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Ustekinumab; Vedolizumab; anti-TNF; CRP; calprotectin; cohort
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three blood samples of 4 ml, one stool sample of 50 mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Ustekinumab: Patients presenting an active crohn's disease (HBI score ≥ 4) with an indication of treatment by ustekinumab because of failure or unacceptable side effects of previous treatments, and who have already been treated by at least one anti TNF The patients must be 18 years old or older.
  Interventions: Biological: Evaluation of biological predictive factors of clinical response to ustekinumab

INTERVENTIONS:
Biological: Evaluation of biological predictive factors of clinical response to ustekinumab — The clinical response is defined as a decrease in the Crohn's Disease Activity Index (CDAI) score ≥ 100 points or a decrease in the HBI score ≥ 3 points.

SUMMARY:
Ustekinumab is a fully human Immune Globulin Gk (IgGk) monoclonal antibody against the common p40 subunit of interleukin-12 and interleukin-23, which are implicated in the pathogenesis of inflammatory bowel disease. Its efficiency to induce and maintain clinical response in patients with anti TNF resistant Crohn's disease has been proved in several clinical trials, and the profile of safety of this treatment was good, but the investigators have few data about biological characteristics of patients treated by Ustekinumab, particularly about ustekinumab through levels and rate of patients developing anti ustekinumab antibodies during the induction and maintenance stages, and no predictive factors of clinical response have been identified yet.

The aim of this study will be to assess the evolution of biological markers of inflammation and ustekinumab trough levels and antibodies, in responders and non responders patients treated by ustekinumab, in order to identify predictive factors of clinical response.

The investigators will perform a prospective observational study, including the patients followed in the University hospital center of Lyon and treated by ustekinumab for a moderate to severe Crohn's disease (with a HBI score≥4 ). All the patients included will have been previously treated by at least one anti TNF and/or Vedolizumab, with specified criteria for a primary non response, a secondary loss of response or unacceptable side effects.

Then, clinical and biological data will be collected for each patient at the inclusion, and then at weeks 4, 8, 16, 24: HBI score, sides effects, extra intestinal manifestations, steroids withdraw, CRP, calprotectin, ustekinumab trough levels and ustekinumab antibodies.

The investigators will compare responding and non responding patients at week 16 (end of the induction period) according to these data.

The hypothesis the investigators state is that an early and significant decrease of the inflammation markers in blood and stools associated with a high ustekinumab through level in blood is associated with a clinical response at week 16 in the patients treated by ustekinumab

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Man or non pregnant woman
* Diagnostic attested of Crohn's disease
* Active Crohn's disease, with HBI score ≥ 4
* Previous treatment by at least one anti TNF and / or vedolizumab,, with primary non response, secondary loss of response or unacceptable side effects
* Formal indication of treatment by ustekinumab
* Patient informed and not opposed to his participation at the study

Exclusion Criteria:

* Pregnancy
* Evolutive cancer
* Evolutive and uncontrolled infection
* Psychiatric pathology that could interfere with the follow-up
* Refusal of the patient

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study is conducted in adults with moderate to severe active Crohn's disease who are resistant to TNF and Vedolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Measurement of serum ustekinumab trough concentrations (expressed in microg/mL) at week 8. | Week 8
  Dosage of ustekinumab through level and ustekinumab antibodies: one 4ml blood sample

SECONDARY OUTCOMES:
Measurement of serum ustekinumab trough concentrations (expressed in microg/mL) at week 4. | Week 4
  Dosage of ustekinumab through level and ustekinumab antibodies: one 4ml blood sample
Measurement of serum ustekinumab trough concentrations (expressed in microg/mL) at week 16. | Week 16
  Dosage of ustekinumab through level and ustekinumab antibodies: one 4ml blood sample
Measurement of serum ustekinumab trough concentrations (expressed in microg/mL) at week 24. | Week 24
  Dosage of ustekinumab through level and ustekinumab antibodies: one 4ml blood sample
Dosage in blood at week 4 | Week 4
  -Inflammation markers are evaluated : Dosage of CRP and leucocytes in blood: two 4ml blood sample
Dosage in blood at week 8 | Week 8
  -Inflammation markers are evaluated : Dosage of CRP and leucocytes in blood: two 4ml blood sample
Dosage in blood at week 16 | Week 16
  -Inflammation markers are evaluated : Dosage of CRP and leucocytes in blood: two 4ml blood sample
Dosage in blood at week 24 | Week 24
  -Inflammation markers are evaluated : Dosage of CRP and leucocytes in blood: two 4ml blood sample
Dosage of calprotectin in stools at week 4 | Week 4
  -Inflammation markers are evaluated : Dosage of calprotectin in stools: one about 50 mg stools sample
Dosage of calprotectin in stools at week 8 | Week 8
  -Inflammation markers are evaluated : Dosage of calprotectin in stools: one about 50 mg stools sample
Dosage of calprotectin in stools at week 16 | Week 16
  -Inflammation markers are evaluated : Dosage of calprotectin in stools: one about 50 mg stools sample
Dosage of calprotectin in stools at week 24 | Week 24
  -Inflammation markers are evaluated : Dosage of calprotectin in stools: one about 50 mg stools sample
Physical evaluation at week 4 | Week 4
  Clinical evaluation is realized by a medical visit with physical examination
Physical evaluation at week 8 | Week 8
  Clinical evaluation is realized by a medical visit with physical examination
Physical evaluation at week 16 | Week 16
  Clinical evaluation is realized by a medical visit with physical examination
Physical evaluation at week 24 | Week 24
  Clinical evaluation is realized by a medical visit with physical examination
Clinical evaluation at week 4 | Week 4
  Clinical evaluation is realized by a medical visit with evaluation of:
  * the efficiency of the treatment: evaluation of well being, abdominal pain, stools numbers per day, presence or not of peri anal lesion, arthralgia, fever
  * the tolerance/potential side effects of the treatment: infections, headache, skin rash, nausea, allergic reaction, or any clinical manifestation that could be imputed to the treatment
Clinical evaluation at week 8 | Week 8
  Clinical evaluation is realized by a medical visit with evaluation of:
  * the efficiency of the treatment: evaluation of well being, abdominal pain, stools numbers per day, presence or not of peri anal lesion, arthralgia, fever
  * the tolerance/potential side effects of the treatment: infections, headache, skin rash, nausea, allergic reaction, or any clinical manifestation that could be imputed to the treatment
Clinical evaluation at week 16 | Week 16
  Clinical evaluation is realized by a medical visit with evaluation of:
  * the efficiency of the treatment: evaluation of well being, abdominal pain, stools numbers per day, presence or not of peri anal lesion, arthralgia, fever
  * the tolerance/potential side effects of the treatment: infections, headache, skin rash, nausea, allergic reaction, or any clinical manifestation that could be imputed to the treatment
Clinical evaluation at week 24 | Week 24
  Clinical evaluation is realized by a medical visit with evaluation of:
  * the efficiency of the treatment: evaluation of well being, abdominal pain, stools numbers per day, presence or not of peri anal lesion, arthralgia, fever
  * the tolerance/potential side effects of the treatment: infections, headache, skin rash, nausea, allergic reaction, or any clinical manifestation that could be imputed to the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Lyon Sud, Pierre-Bénite, France